CLINICAL TRIAL: NCT04735120
Title: Effect of Laser Activation on the Intraoperative and Post-treatment Pain in Single Visit Root Canal Treatment for Mandibular Molar Teeth With Acute Irreversible Pulpitis
Brief Title: Laser Activation in Reducing Pain During and After Root Canal Treatment for Painful Lower Molar Teeth.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSI College of Dental Sciences and Research, Madurai (Other)
Responsible Party: Principal Investigator, Dr SUBASHRI V, Principal investigator, CSI College of Dental Sciences and Research, Madurai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSICDSR
Record Dates: First submitted 2021-01-26; First posted 2021-02-02 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Decayed Teeth
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser to reduce pain intraoperatively and post operatively (Experimental): Diode lasers are used to assess its efficacy in reducing intraoperative and postoperative pain following root canal treatment in mandibular molar teeth with acute irreversible pulpitis
  Interventions: Device: iLASE DIODE LASERS

INTERVENTIONS:
Device: iLASE DIODE LASERS — 940nm diode laser with 1.5 watts activated in a continuous mode and applied on to the canal orifices during root canal treatment to reduce intraoperative pain and further its effect on post operative pain is assessed

SUMMARY:
Effectiveness of lasers in reducing pain during and after root canal treatment for mandibular molar teeth affected with acute irreversible pulpitis.

DETAILED DESCRIPTION:
AIM : To assess the intraoperative and postoperative pain incidence for single visit root canal treatment for mandibular molar teeth with acute irreversible pulpitis following laser activation.

MATERIALS AND METHODS: The study will account the patients who are referred to the Department of Endodontics,both male and female patients,with pain due to acute irreversible pulpitis from carious mandibular first and second molar teeth requiring root canal treatment. Subjects of age 13 to 70 years who met the inclusion criteria and responded positively to cold test will be included in the study.

Single visit root canal treatment with 2.5 mL of 2% lignocaine containing 1:80,000 adrenaline for an inferior alveolar block injection will be administered for each individual. After achieving anesthesia, patients who exhibit pain following access opening will be subjected to diode laser application on the pulp canal orifices. With regard to intraoperative pain, pre laser and post laser intraoperative pain incidence will be recorded. Once when the intraoperative pain incidence is reduced, patients will be reassessed for the need of additional anesthesia. If fully anesthetised, root canal procedure will be completed. Preoperative, intraoperative( before and laser application) pulse rate will also be measured. The levels of preoperative and post-operative pain at 24 hrs and 48 hrs for each patient will be recorded using a 10-point visual analog scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Patients with painful mandibular molar teeth due to caries with no history of medication intake before 7 days prior to root canal treatment
* Patients who respond exaggerated pain with or without lingering response on cold test

Exclusion Criteria:

* Patients who do not have pain upon access opening following local anesthesia administration
* Teeth with poor periodontal or restorative prognosis,
* Patients with serious systemic ailments or conditions hindering single visit root canal treatment
* patients not willing to participate in the post operative recall evaluation
* Teeth with anatomic variations and
* Allergic patients are excluded

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in intraoperative pain measured using visual analog scale during root canal treatment following laser application | procedure (during root canal treatment)
  Change in pain is assessed in 10 point visual analog scale (VAS) before and after laser application.

SECONDARY OUTCOMES:
Change in postoperative pain measured using visual analog scale after root canal treatment | 48 hours
  change in post-operative pain following laser application is assessed using 10 point visual analog scale (VAS) over phone call.

CONTACTS AND LOCATIONS:
Locations (1):
- Csi College of Dental Sciences and Research, Madurai, India

IPD SHARING:
Plan to Share IPD: No